CLINICAL TRIAL: NCT02987543
Title: A Phase III, Open Label, Randomized Study to Assess the Efficacy and Safety of Olaparib (Lynparza™) Versus Enzalutamide or Abiraterone Acetate in Men With Metastatic Castration-Resistant Prostate Cancer Who Have Failed Prior Treatment With a New Hormonal Agent and Have Homologous Recombination Repair Gene Mutations (PROfound)
Brief Title: Study of Olaparib (Lynparza™) Versus Enzalutamide or Abiraterone Acetate in Men With Metastatic Castration-Resistant Prostate Cancer (PROfound Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Foundation Medicine (Industry); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D081DC00007; 2016-000300-28 (EudraCT Number)
Record Dates: First submitted 2016-11-15; First posted 2016-12-09 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer (mCRPC); homologous recombination repair (HRR)
MeSH Terms: interventions — olaparib; enzalutamide; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olaparib (Experimental): Olaparib is available as a film-coated tablet containing 150 mg or 100 mg of olaparib. Subjects will be administered study treatment orally at a dose of 300 mg twice daily (bid). The planned dose of 300 mg bid will be made up of two x 150 mg tablets twice daily, with 100 mg tablets used to manage dose reductions
  Interventions: Drug: olaparib
- Enzalutamide OR abiraterone acetate (Active Comparator): Enzalutamide:
  Enzalutamide is available as capsules or tablets containing 40 mg of enzalutamide. Subjects will be administered study treatment orally at a dose of 160 mg once daily.
  Abiraterone acetate with prednisone: Abiraterone acetate is available as tablets containing 250 mg or 500 mg of abiraterone acetate. Subjects will be administered study treatment orally at a dose of 1,000 mg once daily in combination with prednisone 5 mg administered twice daily orally. Prednisolone is permitted for use instead of prednisone if necessary.
  Interventions: Drug: enzalutamide; Drug: abiraterone acetate

INTERVENTIONS:
Drug: olaparib — 300 mg (2x 150 mg tablets) twice daily
  Other Names: Lynparza
  Arms: Olaparib
Drug: enzalutamide — 160 mg (4 x 40 mg capsules) once daily
  Other Names: XTANDI
  Arms: Enzalutamide OR abiraterone acetate
Drug: abiraterone acetate — 1,000 mg (4 x 250 mg tablets) once daily
  Other Names: ZYTIGA
  Arms: Enzalutamide OR abiraterone acetate
Drug: abiraterone acetate — 1,000 mg (2 x 500 mg tablets) once daily
  Other Names: ZYTIGA
  Arms: Enzalutamide OR abiraterone acetate
Drug: enzalutamide — 160 mg (4 x 40 mg tablets) once daily
  Other Names: XTANDI
  Arms: Enzalutamide OR abiraterone acetate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of olaparib versus enzalutamide or abiraterone acetate in subjects with metastatic castration-resistant prostate cancer who have failed prior treatment with a new hormonal agent and have homologous recombination repair gene mutations.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open-label, phase 3 trial evaluating the efficacy and safety of olaparib versus enzalutamide or abiraterone in subjects with metastatic castration-resistant prostate cancer (mCRPC) who have failed prior treatment with a new hormonal agent (NHA) and have a qualifying tumor mutation in one of 15 genes involved in the homologous recombination repair (HRR) pathway. Subjects will be divided into two cohorts based on HRR gene mutation status.

Approximately 340 subjects will be randomized 2:1 (olaparib : investigator choice of enzalutamide or abiraterone acetate) into the trial.

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed diagnosis of prostate cancer.
2. Documented evidence of metastatic castration resistant prostate cancer (mCRPC).
3. Subjects must have progressed on prior new hormonal agent (e.g. abiraterone acetate and/or enzalutamide) for the treatment of metastatic prostate cancer and/or CRPC .
4. Ongoing therapy with LHRH analog or bilateral orchiectomy.
5. Radiographic progression at study entry while on androgen deprivation therapy (or after bilateral orchiectomy).
6. Qualifying HRR mutation in tumor tissue.

Exclusion criteria

1. Any previous treatment with PARP inhibitor, including olaparib.
2. Subjects who have any previous treatment with DNA-damaging cytotoxic chemotherapy, except if for non-prostate cancer indication and last dose > 5 years prior to randomization.
3. Other malignancy (including MDS and MGUS) within the last 5 years except: adequately treated non-melanoma skin cancer or other solid tumors curatively treated with no evidence of disease for ≥5 years.
4. Subjects with known brain metastases.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, M.D., Ph.D., Principal Investigator — The Institute of Cancer Research, United Kingdom; Maha Hussain, M.D., FACP, FASCO, Principal Investigator — Northwestern University, United States of America
Locations (177):
- United States (33):
  - Research Site, Anchorage, Alaska
  - Research Site, Tucson, Arizona
  - Research Site, Duarte, California
  - Research Site, San Diego, California
  - Research Site, Santa Barbara, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Jeffersonville, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Springfield, Oregon
  - Research Site, Tualatin, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Spokane, Washington
  - Research Site, Wheeling, West Virginia
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, La Rioja
  - Research Site, Rosario
- Australia (10):
  - Research Site, Adelaide
  - Research Site, Box Hill
  - Research Site, Clayton
  - Research Site, Greenslopes
  - Research Site, Herston
  - Research Site, Macquarie University
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Randwick
  - Research Site, Waratah
- Austria (4):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Brazil (12):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Research Site, Odense C, Denmark
- France (13):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (15):
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bremen
  - Research Site, Cologne
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Holzminden
  - Research Site, Jena
  - Research Site, Magdeburg
  - Research Site, Nuremberg
  - Research Site, Nürtingen
  - Research Site, Tübingen
  - Research Site, Wuppertal
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Ẕerifin
- Italy (9):
  - Research Site, Ancona
  - Research Site, Arezzo
  - Research Site, Bari
  - Research Site, Brescia
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Trento
- Japan (26):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Kanazawa
  - Research Site, Kashihara-shi
  - Research Site, Kashiwa
  - Research Site, Kawagoe-shi
  - Research Site, Kita-gun
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsuyama
  - Research Site, Minatoku
  - Research Site, Mitaka-shi
  - Research Site, Miyazaki
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakura-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Hilversum
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Tilburg
  - Research Site, Zwolle
- Research Site, Lørenskog, Norway
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Seoul
- Spain (5):
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Seville
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Solna
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Karşıyaka
- United Kingdom (4):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Romford
  - Research Site, Sutton

REFERENCES:
- [Derived] Mateo J, de Bono JS, Fizazi K, Saad F, Shore N, Sandhu S, Chi KN, Agarwal N, Olmos D, Thiery-Vuillemin A, Ozguroglu M, Mehra N, Matsubara N, Young Joung J, Padua C, Korbenfeld E, Kang J, Marshall H, Lai Z, Barnicle A, Poehlein C, Lukashchuk N, Hussain M. Olaparib for the Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer and Alterations in BRCA1 and/or BRCA2 in the PROfound Trial. J Clin Oncol. 2024 Feb 10;42(5):571-583. doi: 10.1200/JCO.23.00339. Epub 2023 Nov 14. PMID 37963304
- [Derived] Roubaud G, Ozguroglu M, Penel N, Matsubara N, Mehra N, Kolinsky MP, Procopio G, Feyerabend S, Joung JY, Gravis G, Nishimura K, Gedye C, Padua C, Shore N, Thiery-Vuillemin A, Saad F, van Alphen R, Carducci MA, Desai C, Brickel N, Poehlein C, Del Rosario P, Fizazi K. Olaparib tolerability and common adverse-event management in patients with metastatic castration-resistant prostate cancer: Further analyses from the PROfound study. Eur J Cancer. 2022 Jul;170:73-84. doi: 10.1016/j.ejca.2022.04.016. Epub 2022 May 19. PMID 35598359
- [Derived] Matsubara N, Nishimura K, Kawakami S, Joung JY, Uemura H, Goto T, Kwon TG, Sugimoto M, Kato M, Wang SS, Pang ST, Chen CH, Fujita T, Nii M, Shen L, Dujka M, Hussain M, de Bono J. Olaparib in patients with mCRPC with homologous recombination repair gene alterations: PROfound Asian subset analysis. Jpn J Clin Oncol. 2022 May 5;52(5):441-448. doi: 10.1093/jjco/hyac015. PMID 35229141
- [Derived] Thiery-Vuillemin A, de Bono J, Hussain M, Roubaud G, Procopio G, Shore N, Fizazi K, Dos Anjos G, Gravis G, Joung JY, Matsubara N, Castellano D, Degboe A, Gresty C, Kang J, Allen A, Poehlein C, Saad F. Pain and health-related quality of life with olaparib versus physician's choice of next-generation hormonal drug in patients with metastatic castration-resistant prostate cancer with homologous recombination repair gene alterations (PROfound): an open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Mar;23(3):393-405. doi: 10.1016/S1470-2045(22)00017-1. Epub 2022 Feb 11. PMID 35157830
- [Derived] Hussain M, Corcoran C, Sibilla C, Fizazi K, Saad F, Shore N, Sandhu S, Mateo J, Olmos D, Mehra N, Kolinsky MP, Roubaud G, Ozguroglu M, Matsubara N, Gedye C, Choi YD, Padua C, Kohlmann A, Huisden R, Elvin JA, Kang J, Adelman CA, Allen A, Poehlein C, de Bono J. Tumor Genomic Testing for >4,000 Men with Metastatic Castration-resistant Prostate Cancer in the Phase III Trial PROfound (Olaparib). Clin Cancer Res. 2022 Apr 14;28(8):1518-1530. doi: 10.1158/1078-0432.CCR-21-3940. PMID 35091440
- [Derived] Hussain M, Mateo J, Fizazi K, Saad F, Shore N, Sandhu S, Chi KN, Sartor O, Agarwal N, Olmos D, Thiery-Vuillemin A, Twardowski P, Roubaud G, Ozguroglu M, Kang J, Burgents J, Gresty C, Corcoran C, Adelman CA, de Bono J; PROfound Trial Investigators. Survival with Olaparib in Metastatic Castration-Resistant Prostate Cancer. N Engl J Med. 2020 Dec 10;383(24):2345-2357. doi: 10.1056/NEJMoa2022485. Epub 2020 Sep 20. PMID 32955174
- [Derived] de Bono J, Mateo J, Fizazi K, Saad F, Shore N, Sandhu S, Chi KN, Sartor O, Agarwal N, Olmos D, Thiery-Vuillemin A, Twardowski P, Mehra N, Goessl C, Kang J, Burgents J, Wu W, Kohlmann A, Adelman CA, Hussain M. Olaparib for Metastatic Castration-Resistant Prostate Cancer. N Engl J Med. 2020 May 28;382(22):2091-2102. doi: 10.1056/NEJMoa1911440. Epub 2020 Apr 28. PMID 32343890
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081DC00007&attachmentIdentifier=fe1712ee-5e58-4f7d-a072-3044f698908d&fileName=D081DC00007_CSP_redacted.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081DC00007&attachmentIdentifier=441f6e9d-6f12-410a-9352-dca653de8d9c&fileName=D081DC00007_SAP_redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081DC00007&attachmentIdentifier=cedcfc75-9a55-4974-b756-654ad809ea1b&fileName=d081dc00007-addendum-2-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were divided into two cohorts based on HRR gene mutation status. Subjects with mutations in either BRCA1, BRCA2, or ATM are in Cohort A whereas subjects with mutations among 12 other genes involved in the HRR pathway (BARD1, BRIP1, CDK12, CHEK1,CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, or RAD54L) are in Cohort B.
Groups:
- Cohort A Olaparib 300mg bd; Cohort B Olaparib 300mg bd: 2x150mg film-coated tablets
- Cohort A Investigators Choice of NHA; Cohort B Investigators Choice of NHA: either enzalutamide capsules (160 mg od) or abiraterone acetate tablets (1,000 mg od with 5 mg bid prednisone)
Period: Overall Study
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA | Cohort B Olaparib 300mg bd | Cohort B Investigators Choice of NHA
Started | 162 | 83 | 94 | 48
Completed | 0 | 0 | 0 | 0
Not Completed | 162 | 83 | 94 | 48
Not completed — Ongoing study at data cut off | 49 | 21 | 19 | 12
Not completed — Death | 88 | 54 | 67 | 28
Not completed — Lost to Follow-up | 3 | 0 | 1 | 0
Not completed — Screen failure | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 21 | 7 | 7 | 6
Not completed — Study terminated by sponsor | 1 | 0 | 0 | 0
Not completed — Investigator decision | 0 | 1 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA | Cohort B Olaparib 300mg bd | Cohort B Investigators Choice of NHA | Total
Number analyzed (Participants) | 162 | 83 | 94 | 48 | 387
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (8.23) | 68.1 (7.36) | 69.2 (8.79) | 70.3 (7.83) | 68.6 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 162 | 83 | 94 | 48 | 387
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 109 | 55 | 54 | 30 | 248
  Black or African American | 2 | 1 | 5 | 0 | 8
  Asian | 43 | 19 | 26 | 17 | 105
  Other | 1 | 1 | 1 | 0 | 3
  Missing | 7 | 7 | 8 | 1 | 23

OUTCOME MEASURES:

1. Secondary Outcome: Confirmed Objective Response Rate (ORR) by Blinded Independent Central Review (BICR) - Cohort A Only
Description: ORR is the percentage of patients with at least one visit response of Complete response (CR) or Partial response (PR), in their soft tissue disease assessed by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), in the absence of progression on bone scan assessed by Prostate Cancer Working Group 3 (PCWG3)). Per RECIST v1.1, CR=Disappearance of all target lesions; PR = >=30% decrease in the sum of diameters of target lesions; For each treatment group, ORR is the number of patients with a CR and PR.
Time Frame: Tumor assessments every 8 weeks from randomisation until radiographic progression assessed by BICR (median duration of treatment of 7 and 4 months for Olaparib and Investigators Choice of NHA respectively).
Population: Evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA
Number analyzed (Participants) | 84 | 43
Participants
  Response | 28 | 1
  No response | 56 | 42
Statistical Analysis 1: Comparison: Cohort A Olaparib 300mg bd vs Cohort A Investigators Choice of NHA; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 20.86, 95% CI 2-sided [4.18 to 379.18]

2. Secondary Outcome: Radiological Progression Free Survival (rPFS) by Blinded Independent Central Review (BICR) - Cohort A+B
Description: The time from randomisation until the date of objective radiological disease progression (by RECIST 1.1 and Prostate Cancer Working Group 3 (PGWG-3)) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from randomised therapy or received another anti-cancer therapy prior to progression.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA
Number analyzed (Participants) | 256 | 131
Months | 5.82 [5.52 to 7.36] | 3.52 [2.2 to 3.65]
Statistical Analysis 1: Comparison: Cohort A Olaparib 300mg bd vs Cohort A Investigators Choice of NHA; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.38 to 0.63]

3. Secondary Outcome: Time to Pain Progression - Cohort A Only
Description: Time from randomisation to time point at which worsening in pain is observed (ie date of pain progression - date of randomisation + 1). Based on average Brief Pain Inventory - short form (BPI-SF) worst pain [Item 3] and Analgesic Quantification Algorithm [AQA] score.
Time Frame: Every 4 weeks from randomisation (for 7 consecutive days) throughout the study (median duration of treatment of 7 and 4 months for Olaparib and Investigators Choice of NHA respectively).
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA
Number analyzed (Participants) | 162 | 83
Months | NA [NA to NA] — NA - Not calculated, estimates cannot be calculated due to too few events. | 9.92 [5.39 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: Cohort A Olaparib 300mg bd vs Cohort A Investigators Choice of NHA; Test type: Superiority; p = 0.0192, Regression, Cox; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.22 to 0.91]

4. Secondary Outcome: Overall Survival (OS) - Cohort A Only
Description: Number of Participants with Overall Survival (OS) - Cohort A only.
Time Frame: Approximately 35 months after the first patient was randomised.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA
Number analyzed (Participants) | 162 | 83
Participants
  Died | 91 | 57
  Alive at data cut-off | 49 | 21
  Terminated prior to death (withdrawn consent) | 22 | 5
Statistical Analysis 1: Comparison: Cohort A Olaparib 300mg bd vs Cohort A Investigators Choice of NHA; Test type: Superiority; p = 0.0175, Regression, Cox — 2-sided p-value; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.50 to 0.97]

5. Primary Outcome: Radiological Progression Free Survival (rPFS) by Blinded Independent Central Review (BICR) - Cohort A Only
Description: The time from randomisation until the date of objective radiological disease progression (determined by RECIST 1.1 (soft tissue) and Prostate Cancer Working Group 3 (PCWG-3) (bone)) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from randomised therapy or received another anti-cancer therapy prior to progression. Progression is defined using (i) Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for soft tissue, as a >=20% increase in the sum of diameters of target lesions and an absolute increase of >=5mm taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters; (ii) Prostate Cancer Working Group 3 (PGWG-3) for bone as >= 2 new bone lesions on the 1st week 8 scan compared to baseline. The confirmatory scan, >=6 weeks later, must show >=2 more new bone lesions (for a total of >=4 new bone lesions since baseline).
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A Olaparib 300mg bd | Cohort A Investigators Choice of NHA
Number analyzed (Participants) | 162 | 83
Months | 7.39 [6.24 to 9.33] | 3.55 [1.91 to 3.71]
Statistical Analysis 1: Comparison: Cohort A Olaparib 300mg bd vs Cohort A Investigators Choice of NHA; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.25 to 0.47]

ADVERSE EVENTS:
Time Frame: From the time of signature of informed consent throughout the treatment period (median duration of treatment of 7.5 and 3.9 months for Olaparib and Investigators Choice of NHA respectively) up to and including the 30-day follow-up period
Description: There were 131 subjects randomised to the Investigators Choice of NHA treatment group (Full Analysis Set), however 1 of these subjects did not receive treatment (resulting in 130 in the Safety Analysis Set). Hence, for the Investigators Choice of NHA, the Total number at risk for all-cause mortality = 131 while the Total # at Risk by any Serious Adverse Event = 130 and the Total # at Risk by any Other Adverse Event = 130.
Groups:
- Cohort A+B Olaparib 300mg bd: 2x150mg film-coated tablets
- Cohort A+B Investigators Choice of NHA: either enzalutamide capsules (160 mg od) or abiraterone acetate tablets (1,000 mg od with 5 mg bid prednisone)
Arm/Group | Cohort A+B Olaparib 300mg bd | Cohort A+B Investigators Choice of NHA
All-Cause Mortality (participants affected / at risk) | 160/256 | 88/131
Serious Adverse Events (participants affected / at risk) | 94/256 | 39/130
Other Adverse Events (participants affected / at risk) | 241/256 | 112/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A+B Olaparib 300mg bd (N=256) | Cohort A+B Investigators Choice of NHA (N=130)
Anaemia (Blood and lymphatic system disorders) | 23 (24) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stress ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 4 (4) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (3)
Sudden death (General disorders) | 1 (1) | 0 (0)
Budd-Chiari syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 11 (13) | 4 (4)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ballismus (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumoni (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A+B Olaparib 300mg bd (N=256) | Cohort A+B Investigators Choice of NHA (N=130)
Anaemia (Blood and lymphatic system disorders) | 110 (154) | 20 (23)
Constipation (Gastrointestinal disorders) | 49 (52) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 54 (71) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 20 (23) | 3 (3)
Nausea (Gastrointestinal disorders) | 109 (136) | 26 (28)
Vomiting (Gastrointestinal disorders) | 49 (82) | 17 (19)
Asthenia (General disorders) | 37 (54) | 18 (19)
Fatigue (General disorders) | 68 (71) | 28 (28)
Oedema peripheral (General disorders) | 34 (36) | 10 (10)
Pyrexia (General disorders) | 15 (16) | 4 (4)
Urinary tract infection (Infections and infestations) | 18 (22) | 12 (15)
Weight decreased (Investigations) | 21 (21) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 78 (88) | 24 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (26) | 14 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (44) | 17 (18)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 6 (6)
Dizziness (Nervous system disorders) | 17 (18) | 5 (5)
Dysgeusia (Nervous system disorders) | 18 (20) | 2 (2)
Headache (Nervous system disorders) | 16 (29) | 3 (3)
Insomnia (Psychiatric disorders) | 14 (14) | 4 (4)
Haematuria (Renal and urinary disorders) | 6 (7) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (32) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 13 (15) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 13 (16) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (22) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 13 (14) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (18) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT02987543/Prot_005.pdf
  • Statistical Analysis Plan (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT02987543/SAP_015.pdf